CLINICAL TRIAL: NCT01647412
Title: Growth Hormone and Nutrition Therapy in Juvenile Crohn's Disease, a Randomized Clinical Trial
Brief Title: Growth Hormone and Exclusion Diet Therapy in Juvenile Crohn's Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left the institution
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAJ8306
Record Dates: First submitted 2012-07-19; First posted 2012-07-23 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; Inflammatory Bowel Disease; Growth Hormone; Nutraceuticals
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — Growth Hormone; BID protein, human; Fish Oils; Iron; Geritol; Elimination Diets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Growth Hormone, Exclusion Diet, and Nutraceutical therapy (Active Comparator): The experimental group will receive the exclusion diet and nutraceutical therapy (DNT) and daily subcutaneously administered recombinant human growth hormone (rhGH) for the first 26 weeks. After 26 weeks this group will continue on the exclusion diet nutraceutical therapy for the remaining 26 weeks of the study.
  Interventions: Drug: Growth Hormone; Dietary Supplement: Nutraceutical Combination; Other: Exclusion Diet
- rhGH placebo, Exclusion diet, and nutraceutical therapy (Placebo Comparator): The experimental group will receive the exclusion diet and nutraceutical therapy (DNT) and daily subcutaneously administered placebo injections for the first 26 weeks. After 26 weeks this group will continue on the exclusion diet and nutraceutical therapy for the remaining 26 weeks of the study.
  Interventions: Dietary Supplement: Nutraceutical Combination; Other: Exclusion Diet; Other: Placebo Growth Hormone

INTERVENTIONS:
Drug: Growth Hormone — Humatrope will be administered daily to patients in a dose of .18-.20 mg/kg/week.
  Arms: Growth Hormone, Exclusion Diet, and Nutraceutical therapy
Dietary Supplement: Nutraceutical Combination
  Other Names: Jarrow Curcumin oral capsule bid; Jarrow Max DHA (Fish oil) oral capsule daily; Culturelle Probiotics oral capsule tw; Intestive oral capsule bid; Nutrient 950 without Iron (Multivitamin) oral capsule daily
Other: Exclusion Diet — Patients on the exclusion diet will adhere from consumption of all grain, corn, dairy, and carrageenan containing products.
Other: Placebo Growth Hormone
  Arms: rhGH placebo, Exclusion diet, and nutraceutical therapy

SUMMARY:
Of the estimated one million Americans with inflammatory bowel disease (IBD), approximately 20-30% develop this condition during childhood or adolescence, most of whom have Crohn's disease (CD). It appears that some individuals are genetically susceptible to certain nutrients, causing inflammation and disturbance of their immune system, as well as disruption of the intestinal barrier. This leads to malnutrition and inhibited growth, with many patients experiencing intense abdominal pain and diarrhea.

Most physicians treat the disease with drugs that suppress the immune system and decrease the inflammatory process. Although these drugs frequently induce remission, most patients experience a subsequent return of symptoms and fail to catch up on their growth. Additionally, serious side effects are associated with these drugs.

Individuals genetically prone to CD are believed to have a leaky gut that allows substances to pass through the intestinal wall and react with the underlying immune system. Furthermore, those nutrients that are toxic to these individuals pass through the decreased intestinal barrier triggering an extreme immune response. Nutrients that have been implicated include grains, except rice, dairy products, and any food containing carrageenan. Excluding these nutrients from the diet has been shown to beneficial for CD patients. Certain nutraceuticals, such as curcumin and omega-3 fatty acids, have been shown to provide anti-inflammatory effects in IBD patients. In addition, the administration growth hormone (GH), has been shown to alleviate symptoms, by enhancing the repair of the intestinal epithelium, preventing toxic antigens from reaching the underlying lamina propria.

Previous studies and case reports provide incomplete evidence that exclusion diet with nutraceuticals (DNT) and GH lead to sustained long term remission in juvenile CD, discontinuation of other CD drugs, and catch up growth. This study is designed to test this hypothesis. Patients in the treatment group will be treated with DNT and GH, while continuing to receive medications from their physician while the control group will receive DNT, placebo injections instead of GH. We predict that the treatment group will show greater improvement than the control group.

DETAILED DESCRIPTION:
The most widely held hypothesis regarding the pathogenesis of inflammatory bowel disease (IBD) is that overly aggressive acquired immune responses to a subset of commensal enteric bacteria develop in genetically susceptible hosts. In an attempt to avoid disease progression, patients are treated with anti-inflammatory, immunomodulatory and monoclonal antibody drugs, which frequently produce remissions. However, these drugs usually fail to achieve long-term, sustained remission or reversal of growth failure, and are associated with serious side effects. Recently, intestinal barrier dysfunction has been implicated in an alternative 3-step model of IBD pathogenesis.

The investigators hypothesize that the exclusion diet and nutraceutical therapy (DNT) will decrease the production of toxic antigens in the gut and that reactive human growth hormone (rhGH) will reduce the passage of the remaining toxic antigens to the underlying mucosal immune system by promoting the maintenance of the intestinal barrier and accelerating the restitution of the intestinal epithelial lining.

The following study will test whether the the 3-step model is accurate, and whether rhGH and DNT will induce sustained remission in juvenile CD patients.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent
* Age 10-17 years
* Diagnosis of CD as determined by standard clinical, radiological, and pathological criteria
* Clinical evidence of CD for more than 2 years
* Moderate to severely active CD, as defined by a PCDAI score > 30 and < 65
* May continue use of aminosalicylates, antibiotics, immunomodulators, including azathioprine, 6-mercaptopurine and methotrexate, as well as the monoclonal antibody drug, infliximab, if prescribed for at least 4 months and receiving stable doses for at least 2 months prior to baseline visit
* May continue the use of prednisone if prescribed for at least 6 weeks prior to baseline visit
* Meets the following hematological and biochemical requirements:

  * HGB > 8.5 g/dl
  * WBC > 3.5 x 109/L
  * Neut. > 1.5 x 109
  * Plats > 100 x 109/L
  * SGOT & Alk Phos not > 2 times the upper limit of normal

Exclusion Criteria:

* Acute critical illness
* Acute, chronic, or latent infection
* Active neoplasia and/or history of neoplastic disease of any origin other than basal cell carcinoma that has been removed
* Evidence of a systemic disorder unrelated to CD involving hepatic, gastrointestinal, pulmonary, cardiac, renal, hematologic, endocrine, central or peripheral nervous systems
* Use of parenteral corticosteroids or corticotrophin within 2 months of baseline visit
* Use of another investigational agent within 3 months of baseline visit
* Long-term anti-coagulant therapy or use of any anti-coagulant medication, including NSAIDs or ASA, within 2 weeks of screening visit
* Pregnancy (positive pregnancy test)
* Positive stool culture for enteric pathogens, pathogenic ova, parasites or clostridium difficile toxin
* Any condition that the investigator believes would pose significant harm to the subject if the investigational therapy were initiated
* Diagnosis of short bowel syndrome and also on TPN
* Presence of an ostomy, symptomatic stenosis or ileal stricture, or severe intestinal stricture, proctocolectomy, total colectomy or stoma
* Patients in imminent need of surgery due to active gastrointestinal bleeding fixed stenosis, intermittent obstruction or obstructive event within 2 months prior to screening.
* Patients who underwent CD surgery within 2 months of screening

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2012-03

PRIMARY OUTCOMES:
Proportion of Patients in remission | 26 weeks and 52 weeks
  The proportion of patients in remission in each group will be assessed and compared to each other in order to demonstrate efficacy of treatment. Remission will be assessed by a change in the patients PCDAI score to below 10.

SECONDARY OUTCOMES:
Bone Mineral Density (BMD) | Baseline and 52 weeks
  BMD of the hip and spine will be obtained by dual-emission x-ray absorptiometry (DXA) at the baseline visit and week 52.

CONTACTS AND LOCATIONS:
Overall Officials: Alfred E Slonim, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Department of Clinical Genetics, New York, New York, United States